CLINICAL TRIAL: NCT02446197
Title: Self Directed Stations for the Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 014-203
Record Dates: First submitted 2015-02-19; First posted 2015-05-18 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Directed Exercise Group (Experimental): Participants will complete a combination of PT and OT activities that will be individually prescribed based on an evaluation by the therapy team completed pre-intervention. The activities will be added to the comprehensive inpatient rehabilitation program.
  Interventions: Other: Patient Directed Exercise Group
- Standard of care (No Intervention): Standard of care comprehensive inpatient rehabilitation program.

INTERVENTIONS:
Other: Patient Directed Exercise Group — Combination of PT and OT activities that will be individually prescribed based on an evaluation by the therapy team completed pre-intervention. The activities will be added to the comprehensive inpatient rehabilitation program.
  Arms: Patient Directed Exercise Group

SUMMARY:
Early initiation of therapy post stroke has been associated with improved long-term outcomes, and functional activity dose during the first week of inpatient rehabilitation predicts both gait velocity at discharge and length of time to independent walking. The primary study objective is to pilot the feasibility of integrating a patient-directed activity program into inpatient rehabilitation following stroke. The second study objective is to identify if participation in the patient-directed activity program improves functional ability and health related quality of life.

DETAILED DESCRIPTION:
1 BACKGROUND AND RATIONALE

1.1 Background

Due to the high incidence of stroke, increased risk of developing secondary (e.g., pain, depression, urinary tract infections, pressure ulcers, falls, and seizures) and chronic conditions (e.g., second stroke, CVD), high medical costs 1, evolving healthcare system (e.g., reimbursement, length of stay, staffing productivity 2, healthcare professionals are challenged to explore and develop innovative strategies to continue to achieve the best clinical practice and outcomes for patients. Functional activity levels are typically low during inpatient rehabilitation post stroke 3-6, emphasized by King and colleagues 7 who reported that patients post stroke undergoing inpatient rehabilitation spent 76% of their day in their bedroom and 62% being inactive. Consequently, since dose of functional activity (amount of active time and/or quantity of repetitions) is posited to relate to outcomes 8-11, the optimal conditions for inpatient rehabilitation are being questioned. The literature is clear that low functional activity reflects low potential for neuroplasticity. Consequently, novel and feasible methods to provide higher doses of functional activity during inpatient rehabilitation, that realistically considers cost-effectiveness and resource allocation 12, are important to improve functional outcomes post stroke 13.

1.2 Rationale for Protocol

Early initiation of therapy post stroke has been associated with improved long-term outcomes 14, and functional activity dose (e.g., activity time, number of repetitions) during the first week of inpatient rehabilitation predicts both gait velocity at discharge and length of time to independent walking 15. Specifically, patients who completed more than the median number of exercise repetitions (703) during the first week of inpatient rehabilitation experienced quicker recovery of unassisted walking 15. This lack of activity is a significant issue during inpatient rehabilitation and for overall recovery as repetitive task practice is argued to drive neural plasticity following stroke 16,17. Specifically, there is a growing body of evidence indicating that increased functional activity and large volume of practice during inpatient rehabilitation is required to induce improved stretch reflex modulation and increased neuromuscular activation 11, thus leading to meaningful neural adaptations and recovery following stroke 16. However, our current clinical practice of 3-hours of therapy during inpatient rehabilitation (which is standard of care for inpatient rehabilitation hospitals) may not be adequate to facilitate neuroplasticity and achieve optimal functional outcomes 10. This is emphasized by the fact that Medicare beneficiaries with stroke undergoing inpatient rehabilitation experienced shorter LOS, had worsening admission and discharge function, and had fewer community discharges 18. Therefore, our objective in this proposal is to evaluate the feasibility and effectiveness of implementing a novel intervention to facilitate patient-directed activity for individuals undergoing inpatient rehabilitation. The goal of the intervention is to increase repetition, stimulation, attention, and therapeutic activity of the affected extremities and trunk to facilitate improved outcomes following stroke 17,19,20. This will be achieved by adding up to 1.5-hours of daily patient-directed activities into the individuals schedule beyond the 3-hours of therapy provided by clinicians, thus increasing daily therapeutic activity time by up to 50%. The activities will include physical (PT) and occupational therapy (OT) tasks (see table 1 below for more details). The activities are therapeutic in nature, include typical activities that patients would complete during the 3-hours of therapy provided as standard of care, are low intensity, and include activities that involve being seated or prone on a gym mat.

It is important to note that the clinical team at Baylor Institute for Rehabilitation has been implementing up to 1.5-hours of additional daily therapy into standard of care since January 2014. However, to date we have not collected any effectiveness data so the clinical and research team wanted to demonstrate through a research project that the addition of the extra 1.5-hours of daily therapy is beneficial beyond the 3-hours of therapy currently provided as standard of care. Since starting the additional therapy in January 2014 the clinical team has had 25 patients successfully move through rehabilitation and no patients have had any adverse events.

2.1 Primary Objectives

Pilot the feasibility of integrating the novel patient-directed activity program into inpatient rehabilitation following stroke. Based on guidelines for conducting an a priori pilot study we will assess aspects of the process (e.g., eligibility, randomization), resources (e.g., equipment, space), management (e.g., staff capacity for data entry and management), and scientific basis (e.g., sensitive outcome measures) of the intervention. Our working hypothesis is that that the patient-directed activity program will be successfully integrated into patient and clinical schedule.

2.2 Secondary Objectives

To identify if participation in the novel patient-directed activity program improves functional ability and health related quality of life (HRQOL) in patients post stroke. Our working hypothesis is that patients' post stroke that actively participate in the program will manifest significant increases in functional ability and HRQOL at discharge to inpatient rehabilitation and at the follow-up appointment within 6 months of discharge when compared to controls.

3 INVESTIGATIONAL PLAN

3.1 Study Design

We will use a randomized controlled trial and include stroke patients who are undergoing inpatient rehabilitation at Baylor Institute for Rehabilitation (BIR). Participants will be randomized into an experimental (patient-directed station program) or control group (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Safe to be left unsupervised as deemed by therapist or has caregiver present
* Diagnosed with stroke in past six months
* Medically stable as deemed by therapy team
* >3 on FIM comprehension
* Primary diagnosis of stroke (all types)

Exclusion Criteria:

* Pre-morbid developmental disability
* Significant pre-morbid psychological diagnosis or concurrent TBI
* Other cognitive impairment that would prevent participation as determined by the clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Rehabilitation Participation Scale | Daily during inpatient rehab hospitalization, time frame maximum is up to 3 months
  Daily measurements will be recorded during inpatient hospitalization to capture changes in participation between admission and discharge and to calculate sums/averages of participation.

SECONDARY OUTCOMES:
Stroke Rehabilitation Assessment of Movement Measure (STREAM) | Wtihin one week of rehab inpatient admission, within one week of rehab inpatient discharge, at post discharge follow up (3-6 months after inpatient rehab discharge)
WOLF Motor Function Test | Wtihin one week of rehab inpatient admission, within one week of rehab inpatient discharge, at post discharge follow up (3-6 months after inpatient rehab discharge)
Actigraph | Wtihin one week of rehab inpatient admission, within one week of rehab inpatient discharge
Functional Independence Measure | Wtihin one week of rehab inpatient admission, within one week of rehab inpatient discharge, at post discharge follow up (3-6 months after inpatient rehab discharge)
Stroke Impact Scale | Within one week of rehab inpatient discharge, at post discharge follow up (3-6 months after inpatient rehab discharge)
Patient Participation Survey | Within one week of rehab inpatient discharge
Therapist Feasibility Survey | After patient accrual, up to 12 months
  After all patients have been accrued, a one-time feasibility survey will be distributed to treating therapists to assess feasibility with implementing extra physical activity with stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Trammell, PT, Principal Investigator — Physical Therapist
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States